CLINICAL TRIAL: NCT05564013
Title: Developing a Virtual Reality (VR)-Based Prototype for Perioperative Care - a Proof of Concept Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changi General Hospital (Other)
Collaborators: KK Women's and Children's Hospital (KKH) (Unknown)
Responsible Party: Principal Investigator, Lydia Li Weiling, Consultant, Department of Anaesthesia and Surgical Intensive Care, Changi General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIRTUAL02
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Anxiety; Postoperative Pain; Pain, Acute
Keywords: virtual reality; pain management; satisfaction experience
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 - Patient feedback and needs analysis (No Intervention): To facilitate the development of virtual reality application that is suitable for perioperative care management, a survey will be conducted in 100 subjects to gather patient preference and feedback with needs analysis.
- Phase 2 - Evaluation of prototype efficacy (Experimental): Comparison of pre-operative anxiety and post-operative pain in 60 patients before and after intervention using the developed virtual reality application.
  Interventions: Device: Virtual reality

INTERVENTIONS:
Device: Virtual reality — Up to 25 minutes of virtual reality exposure in supine position
  Arms: Phase 2 - Evaluation of prototype efficacy

SUMMARY:
Preoperative anxiety and acute post-operative pain are common and have been associated with the development of chronic post-surgical pain and longer hospitalisation. Pharmacological interventions to combat anxiety and pain come with their attendant adverse effects. Therefore, non-pharmacological strategies- Virtual Reality (VR) has gained popularity to improve overall the perioperative experience for patients.

Our overall aim is to develop and evaluate the use of a VR-based prototype to reduce pre-operative anxiety and post-operative acute pain intensity in our local patient population. Our primary aim is to reduce preoperative anxiety as measured by a reduction in Visual Analogue Score-Anxiety (VAS-A) by a mean of 2.5 points pre-post VR intervention. Our secondary aims are to reduce post-operative acute pain and to achieve more than 50% good to excellent self-reported satisfaction on our VR prototype.

DETAILED DESCRIPTION:
This will be a multi-center, prospective cohort study to be conducted in Changi General Hospital (CGH) and KKH, in collaboration with industry partner, Vue Networks. The patients will provide written informed consent for the study.

Phase 1: To facilitate the development of VR application that is suitable for perioperative care management, a survey will be conducted in 100 subjects (CGH: n=50; KKH: n=50) to gather patient preference and feedback with needs analysis.

The VR application development needs analysis would focus on:

i) instructional module on surgical journey; and ii) mindfulness module with inputs from perspectives of clinical health psychology iii) local relaxation scenarios (e.g. village, botanic gardens, Changi beach, Gardens by the bay); iv) feedback on hardware, i.e., VR headset usability.

Phase 2: The testing of the developed VR application will be performed in 60 subjects (CGH: n=30; KKH: n=30).

The study will utilize Head-Mounted Displays (HMD) such as the PicoG2 4K, the Oculus Go and/or Quest headsets. In immersive VR, high resolution 360-degree video and/or 3D computer graphics are paired with suitable ambience sounds and audio cues to fully immerse the user in the selected environment. The contents comprise a mixture of live-action and/or animation, as well as local settings. The domain components of the VR intervention include:

* VR application for pre-operative anxiety and post-operative acute pain treatment with local context;
* Patient feedback on local scenarios and content of VR and mindfulness;
* Development of VR application: Vue Networks' platform with local and foreign context scenarios, passive and active scenario features, development of mindfulness application, language use for mindfulness application.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21 years old and above and undergoing scheduled surgery;
* American Society of Anesthesiologist physical status I to III, with no visual or hearing impairment; and
* Understands English or Chinese.

Exclusion Criteria:

* Comorbidities affecting usage of virtual reality e.g., giddiness, motion sickness, claustrophobia, stroke, seizure, dementia, transmissible diseases, severe facial eczema; and
* Unable to understand the administered questionnaires.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Pre-operative anxiety | up to 1hour
  Anxiety score - VAS-A (0 to 10; 0-best outcome, 10-worst outcome)

SECONDARY OUTCOMES:
Post-operative pain | up to 1hour
  Pain score - Numerical Rating Scale (0 to 10; 0-best outcome, 10-worst outcome)
User satisfaction | up to 1hour
  Self-reported satisfaction score (0 to 10; 0-worst outcome, 10-best outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Weiling Li, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan JJI, Yeam CT, Kee HM, Tan CW, Sultana R, Sia ATH, Sng BL. The use of pre-operative virtual reality to reduce anxiety in women undergoing gynecological surgeries: a prospective cohort study. BMC Anesthesiol. 2020 Oct 9;20(1):261. doi: 10.1186/s12871-020-01177-6. PMID 33036555
- [Background] Goldman RD, Behboudi A. Virtual reality for intravenous placement in the emergency department-a randomized controlled trial. Eur J Pediatr. 2021 Mar;180(3):725-731. doi: 10.1007/s00431-020-03771-9. Epub 2020 Aug 10. PMID 32779029